CLINICAL TRIAL: NCT03440541
Title: Uses of Gamma Irradiated Amniotic Membrane as an Alternative Method in Psoriasis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Atomic Energy Authority (Other Government)
Responsible Party: Principal Investigator, Nashwa Radwan, Director, Egyptian Atomic Energy Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4102017NCRRT
Record Dates: First submitted 2017-11-29; First posted 2018-02-22 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Psoriasis
Keywords: Amniotic membrane; Psoriasis; Treatment
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treated (Experimental): Patients who received patches of REGE pro on psoriasis lesion weekly for 8 weeks
  Interventions: Combination Product: REGE pro

INTERVENTIONS:
Combination Product: REGE pro — REGE pro is a patch of human amniotic membrane sterilized by gamma radiation

SUMMARY:
Using of human amniotic membrane extra-cellular matrix as a topical treatment for improving Psoriasis Area and Severity Index (PASI).

DETAILED DESCRIPTION:
Human amniotic membrane extra-cellular matrix was purchased from National center for radiation research and technology, Egypt, under commercial name REGE pro gel.

ELIGIBILITY:
Inclusion Criteria:

* patients have psoriasis lesion

Exclusion Criteria:

* must stop other line of treatment

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2015-08-04 (Actual); Primary Completion 2016-02-13 (Actual); Study Completion 2016-04-08 (Actual)

PRIMARY OUTCOMES:
Scaling size decrement | 2 weeks
  REGE pro gel decreased scaling size in patients with sever scales to moderate scale within two weeks, scaling size decrement from moderate to mild within two weeks, and from mild to complete curing within two weeks
Histopathological improvement | 6 weeks
  Two biopsies were taken from each patient before and at the end of the treatment. It was noted that all histological signs as munro's microabscess and the elongation of rete ridges were absent.

SECONDARY OUTCOMES:
Erythema disappearing | 4-6 weeks
  REGE pro gel gradually decreased erythema in patients within 4-6 weeks, these data were collected from applied patients by questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Nashwa K Radwan, PhD, Study Director — NATIONAL CENTER FOR RADIATION RESEARCH AND TECHNOLOGY
Locations (1):
- Amniotic tissue lab, Cairo, Egypt

REFERENCES:
- [Background] Alikarami F, Yari F, Amirizadeh N, Nikougoftar M, Jalili MA. The Immunosuppressive Activity of Amniotic Membrane Mesenchymal Stem Cells on T Lymphocytes. Avicenna J Med Biotechnol. 2015 Jul-Sep;7(3):90-6. PMID 26306147
- [Background] Bata-Csorgo Z, Hammerberg C, Voorhees JJ, Cooper KD. Intralesional T-lymphocyte activation as a mediator of psoriatic epidermal hyperplasia. J Invest Dermatol. 1995 Jul;105(1 Suppl):89S-94S. doi: 10.1111/1523-1747.ep12316121. PMID 7616005
- [Background] Chen CP, Chen YY, Huang JP, Wu YH. The effect of conditioned medium derived from human placental multipotent mesenchymal stromal cells on neutrophils: possible implications for placental infection. Mol Hum Reprod. 2014 Nov;20(11):1117-25. doi: 10.1093/molehr/gau062. Epub 2014 Aug 19. PMID 25140001
- [Background] Gisondi P, Di Mercurio M, Idolazzi L, Girolomoni G. Concept of Remission in Chronic Plaque Psoriasis. J Rheumatol Suppl. 2015 Nov;93:57-60. doi: 10.3899/jrheum.150638. PMID 26523059
- [Background] John T, Foulks GN, John ME, Cheng K, Hu D. Amniotic membrane in the surgical management of acute toxic epidermal necrolysis. Ophthalmology. 2002 Feb;109(2):351-60. doi: 10.1016/s0161-6420(01)00900-9. PMID 11825823
- [Background] Kronsteiner B, Wolbank S, Peterbauer A, Hackl C, Redl H, van Griensven M, Gabriel C. Human mesenchymal stem cells from adipose tissue and amnion influence T-cells depending on stimulation method and presence of other immune cells. Stem Cells Dev. 2011 Dec;20(12):2115-26. doi: 10.1089/scd.2011.0031. Epub 2011 Apr 19. PMID 21381973
- [Background] Li J, Koike-Soko C, Sugimoto J, Yoshida T, Okabe M, Nikaido T. Human Amnion-Derived Stem Cells Have Immunosuppressive Properties on NK Cells and Monocytes. Cell Transplant. 2015;24(10):2065-76. doi: 10.3727/096368914X685230. Epub 2014 Oct 20. PMID 25333453
- [Background] Ma L, Zhou Z, Zhang D, Yang S, Wang J, Xue F, Yang Y, Yang R. Immunosuppressive function of mesenchymal stem cells from human umbilical cord matrix in immune thrombocytopenia patients. Thromb Haemost. 2012 May;107(5):937-50. doi: 10.1160/TH11-08-0596. Epub 2012 Mar 8. PMID 22398715
- [Background] Magatti M, Caruso M, De Munari S, Vertua E, De D, Manuelpillai U, Parolini O. Human Amniotic Membrane-Derived Mesenchymal and Epithelial Cells Exert Different Effects on Monocyte-Derived Dendritic Cell Differentiation and Function. Cell Transplant. 2015;24(9):1733-52. doi: 10.3727/096368914X684033. Epub 2014 Aug 19. PMID 25259480
- [Background] Mahil SK, Capon F, Barker JN. Update on psoriasis immunopathogenesis and targeted immunotherapy. Semin Immunopathol. 2016 Jan;38(1):11-27. doi: 10.1007/s00281-015-0539-8. Epub 2015 Nov 16. PMID 26573299
- [Background] McDonald CA, Payne NL, Sun G, Moussa L, Siatskas C, Lim R, Wallace EM, Jenkin G, Bernard CC. Immunosuppressive potential of human amnion epithelial cells in the treatment of experimental autoimmune encephalomyelitis. J Neuroinflammation. 2015 Jun 3;12:112. doi: 10.1186/s12974-015-0322-8. PMID 26036872
- [Background] Pianta S, Bonassi Signoroni P, Muradore I, Rodrigues MF, Rossi D, Silini A, Parolini O. Amniotic membrane mesenchymal cells-derived factors skew T cell polarization toward Treg and downregulate Th1 and Th17 cells subsets. Stem Cell Rev Rep. 2015 Jun;11(3):394-407. doi: 10.1007/s12015-014-9558-4. PMID 25348066
- [Background] Redondo P, Gimenez de Azcarate A, Marques L, Garcia-Guzman M, Andreu E, Prosper F. Amniotic membrane as a scaffold for melanocyte transplantation in patients with stable vitiligo. Dermatol Res Pract. 2011;2011:532139. doi: 10.1155/2011/532139. Epub 2011 Aug 18. PMID 21869882
- [Background] Yamahara K, Harada K, Ohshima M, Ishikane S, Ohnishi S, Tsuda H, Otani K, Taguchi A, Soma T, Ogawa H, Katsuragi S, Yoshimatsu J, Harada-Shiba M, Kangawa K, Ikeda T. Comparison of angiogenic, cytoprotective, and immunosuppressive properties of human amnion- and chorion-derived mesenchymal stem cells. PLoS One. 2014 Feb 14;9(2):e88319. doi: 10.1371/journal.pone.0088319. eCollection 2014. PMID 24551087